CLINICAL TRIAL: NCT03214458
Title: Tolerance and Acute Effects of Humidified Nasal High-flow With Oxygen (HNHF-O2) on Gas Exchange in Patients Hospitalized With an Acute Exacerbation of COPD
Brief Title: Effects of Nasal High-flow Oxygen in Patients With an Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24408
Record Dates: First submitted 2017-06-19; First posted 2017-07-11 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Therapy; Noninvasive Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nasal high flow with oxygen (Other): During HFNC-oxygen, oxygen will be passed through a heated humidifier (AIRVO-2, Fisher and Paykel Healthcare) and applied continuously through large-bore binasal prongs (Optiflow+ Fisher and Paykel Healthcare), with a gas flow rate of 20-35 liters per minute or as high as the patient will tolerate and an FiO2 to keep Arterial oxygen saturation (SaO2) > 90%. Temperature will be adjusted based on patient's comfort and range from 34-37 degrees based on prior experience.
  Interventions: Device: Nasal high flow

INTERVENTIONS:
Device: Nasal high flow — The AIRVO 2 is for the treatment of spontaneously breathing patients who would benefit from receiving high flow warmed and humidified respiratory gases/

SUMMARY:
The investigators are looking at the effect of humidified nasal high-flow with oxygen (HNHF-O2) on air exchange during exacerbations of COPD. HNHF-O2 therapy may have beneficial effects in patients with severe breathing impairment that results in low oxygen in the blood. Some studies show that patients with low blood oxygen levels who use HFNC oxygen have lower rates of needing mechanical ventilation.

DETAILED DESCRIPTION:
Patients admitted to the hospital with an exacerbation of COPD accompanied by respiratory failure need supplemental oxygen and alleviation of an increased work of breathing. Patients with acute exacerbations of COPD have hypoxemia, hypercapnia and an elevated work of breathing due to increased airways obstruction and hyperinflation. Patient outcomes can be improved by aggressive bronchodilation and systemic corticosteroids, but methods that can augment spontaneous ventilation and decrease the work of breathing can help avoid intubation. High flow nasal cannula (HFNC) has been shown to be useful in patients with severe hypoxemic respiratory failure and those recently extubated from mechanical ventilation. HFNC provides warmed and humidified high flow (10-60L/min) by nasal cannula that allows precise titration of % inspired FiO2 in the air/oxygen blend. The AIRVO 2 device delivers warmed and humidified respiratory gases to spontaneously breathing patients using a humidifier and integrated flow generator. In this study, the air/ oxygen gas blend (20-35L/min) will be administered by the AIRVO 2 HNHF device to achieve an fraction of inspired oxygen (FiO2) > 90% at rest. A potential advantage of the AIRVO 2 HNHF device includes the ability of the device to deliver oxygen that has been warmed and humidified. Also, the high flow rates achieved with this device may reduce the work of breathing. This is an open-labeled pilot study of ten patients to determine the safety and feasibility of using the device in the management of patients with an acute exacerbation of COPD with acute on chronic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 40 years of age or older
* Hospitalized for an acute exacerbation of COPD on the 6th floor of Rock Pavilion (pulmonary inpatient service)
* Smoking history of > 10 pack-years
* PaCO2 ≥ 45 mm Hg
* Able to provide informed consent
* Willing to participate in daily measurements of arterial blood gases, completion of study questionnaires, and other study-related procedures

Exclusion Criteria:

* Upper airway or nasal problems that prohibit the use of humidified high-flow nasal oxygen
* Hemodynamic instability defined as the need for blood pressure or blood volume support to maintain adequate tissue perfusion and oxygenation
* Urgent need for endotracheal intubation
* A do-not-intubate order
* A known diagnosis of obstructive sleep apnea
* Present use of continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BIPAP) therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Ability to maintain oxygen saturation at or above 90% | 3 days
  The need to intensify therapy because HNHF-O2 does not achieve the targeted oxygen saturation of ≥ 90% resulting in the need to intensify respiratory support

SECONDARY OUTCOMES:
Tolerance of HNHF-O2 measured by a 5-point Likert Scale | 3 days
  Likert scale model indicating marked improvement (+2), slight improvement (+1), no change (0), slight deterioration (-1) and marked deterioration (-2) in patient's sensation of shortness of breath.
Tolerance of HNHF-O2 measured by a 100 mm visual analog scale | 3 days
  Discomfort assessed using an unmarked 100 mm visual analogic scale from "no discomfort" to "maximal imaginable discomfort"

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No